CLINICAL TRIAL: NCT04547816
Title: Evaluation of Complex (Physical Therapy and Diet) Treatment of Functional Defecatory Disorders in Females With Pelvic Organ Prolapse
Brief Title: Efficacy of Conservative Treatment of Functional Defecatory Disorders in Females With Pelvic Organ Prolapse
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Federal State Budgetary Scientific Institution "Federal Research Centre of Nutrition, Biotechnology (Other)
Collaborators: State Scientific Centre of Coloproctology, Russian Federation (Other Government); Ministry of Health, Russian Federation (Other Government); Ministry of Science and Higher Education, Russian Federation (Unknown)
Responsible Party: Principal Investigator, Sergey Morozov, MD, PhD, Federal State Budgetary Scientific Institution "Federal Research Centre of Nutrition, Biotechnology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DGH-SSCC1
Record Dates: First submitted 2020-09-01; First posted 2020-09-14 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Pelvic Floor Prolapse; Functional Constipation; Rectocele
Keywords: pelvic floor prolapse; conservative treatment; functional disorders of defecation; rectocele; diet modification; biofeedback therapy; tibial neuromodulation
MeSH Terms: conditions — Rectocele | interventions — Biofeedback, Psychology; Diet Therapy

STUDY DESIGN:
Intervention Model Description: Random assignment to one of the groups depending on the treatment options:
  1. biofeedback and tibial neuromodulation
  2. biofeedback and tibial neuromodulation + pelvic floor muscles training
  3. biofeedback and tibial neuromodulation + pelvic floor muscles training + diet modification
Who Masked: Investigator, Outcomes Assessor
Masking Description: After randomization eligible subjects are to receive one of the treatment option described in the Model Description according to the order placed in a closed envelope which is to be opened by person who perform biofeedback (BFT) and tibial neuromodulation (TNM). The investigator responsible for the study conduction, clinical assessment and high-resolution anorectal manometry measurements is not supposed to get the information about the number of procedures (BFT+TNM; or BFT+TNM + pelvic floor muscles training (PFMT); or BFT+TNM + PFMT + diet modification (DM)) that a certain subject receives
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- biofeedback and tibial neuromodulation (BFB+TNM) (Experimental)
  Interventions: Procedure: Biofeedback therapy; Procedure: Tibial neuromodulation
- BFB+TNM + pelvic floor muscles training (PFMT) (Experimental)
  Interventions: Procedure: Biofeedback therapy; Procedure: Tibial neuromodulation; Behavioral: Pelvic floor muscles training
- BFB+TNM+PFMT+diet modification (Experimental)
  Interventions: Procedure: Biofeedback therapy; Procedure: Tibial neuromodulation; Behavioral: Pelvic floor muscles training; Behavioral: Diet modification

INTERVENTIONS:
Procedure: Biofeedback therapy — Biofeedback therapy is a procedure when the patient is taught to make proper squeezing by adequate increase of intra-abdominal and rectal pressures and relaxation of the muscles of the pelvic floor. This procedure is widely described and is to be performed with the use of devices registered for this purpose Urostim and WPM Solar, MMS, the Netherlands
  Other Names: BFB
Procedure: Tibial neuromodulation — TNM is a standard procedure that is previously described as an effective method to treat functional insufficiency of the anal sphincter. It acts on the lumbosacral nerve plexus with an electric current through the posterior tibial nerve of one of the patient's limbs. For the study purpose a registered device for electric therapy (BioBravo, MTR Plus Vertriebs GmbH, Germany) is to be used.
  Other Names: TNM
Behavioral: Pelvic floor muscles training — PFMT is a complex of 5 exercises aimed to make functional training of pelvic floor muscles. This complex does not require additional equipment. It may be performed at home. The patients will be trained to perform this complex of exercises by a healthcare provider.
  The complex of physical therapy consists of a single basic exercise for training coordinated muscle tension of abdominal wall and relaxation of the pelvic floor muscles, and 4 exercises to increase the contractility of pelvic floor muscles without additional involvement of the muscles of the abdominal wall. This allows to coordinate and consciously control the contraction and relaxation of the pelvic diaphragm. Initial course of training is 10 working days. Than patients continue the intervention for 6 months at home with online monitoring of the correctness and regularity of training.
  Other Names: PFMT
  Arms: BFB+TNM + pelvic floor muscles training (PFMT); BFB+TNM+PFMT+diet modification
Behavioral: Diet modification — Diet modification play an important role in the regulation of colonic transit and defecation. Dietary factors may act through faecal bulk by additional stimulation of mechanoreceptors of the rectum. At the same time, adequate intake of vitamins (for example, B12) may improve electric conductivity of nerves and thus impact the tone of pelvic floor muscles. Among other factors known to affect functional state of pelvic floor muscles and colonic transit are dietary fibers, adequate intake of water, regular meal intake. For the study purposes, it is planned to provide standard recommendation based on the national recommended daily allowances according to patients' sex, age and physical activity level.
  Other Names: DM
  Arms: BFB+TNM+PFMT+diet modification

SUMMARY:
This study is planned to evaluate the efficacy of complex conservative treatment (including tibial neuromodulation, biofeedback therapy, special pelvic floor training and diet modification) in women with pelvic organ prolapse

DETAILED DESCRIPTION:
Pelvic organ prolapse is a condition with impaired anatomic structure, which may result in defecatory disorders and usually considered as an indication for surgery. However, operation is not always possible. Existing data suggest that functional component may also be possible, despite on the anatomic impairment. The aim of the study is to evaluate the effect of complex conservative treatment of functional defecatory disorders in patients with mild to moderate grade of pelvic organ prolapse

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate (signed informed consent form)
* Females with rectocele I-II grade or rectocele I-II grade and internal rectal invagination and functional defecatory disorders (per Rome IV guidelines) confirmed on the basis of complex examination including high-resolution anorectal manometry

Exclusion Criteria:

* rectocele III grade;
* internal genitals prolapse;
* history of abdominal or pelvic surgery that may impact bowel motility (excluding non-complicated appendectomy or laparoscopic cholecystectomy);
* gynecological surgery that may influence sensory or reservoir function of rectum;
* history of major cardiovascular events, or presence of current conditions that in case of participation of the patient in the study may put her at risk of exacerbation or complication;
* start of any new concomitant medication with mechanisms of action that influence rectal motility, sensory function, muscle tone and/or contractility
* inability to understand and/or follow the instructions to perform all the procedures required per protocol
* general condition of the patient that make her ineligible by the discretion of the investigator

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Mean stool frequency | A week
  clinical outcome
Mean stool form value | A week
  clinical outcome, assessed with the use of the Bristol stool scale (BSS)
Mean defecation with difficult bowel emptying | a week
  patient-reported outcome, clinical
Change of KESS scale points | at the end-point, 6 months after enrolment
  A specialized validated questionnaire will be used before treatment and at the end of the study. "Change" is to be assessed as percentage decline from baseline values.
Change in Scale of bowel evacuatory function assessment | at the end-point, 6 months after enrolment
  A specialized validated questionnaire will be used before treatment and at the end of the study. "Change" is to be assessed as percentage decline from baseline v
Average anal resting pressure | at the end-point, 6 months after enrolment
  Values obtained during HR anorectal manometry
Maximum absolute anal squeeze pressure | at the end-point, 6 months after enrolment
  Values obtained during HR anorectal manometry
Average absolute anal squeeze pressure | at the end-point, 6 months after enrolment
  Values obtained during HR anorectal manometry
Average incremental anal squeeze pressure | at the end-point, 6 months after enrolmentat the end-point, 6 months after enrolment
  Values obtained during HR anorectal manometry
Residual push pressure | at the end-point, 6 months after enrolment
  Values obtained during HR anorectal manometry
Push relaxation percentage | at the end-point, 6 months after enrolment
  Values obtained during HR anorectal manometry

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - Federal State Budgetary Scientific Institution "Federal Research Centre of Nutrition, Biotechnology, Moscow
  - Federal Research Center of Coloproctology, Moscow

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: within 2 years after study completion
Access Criteria: per request
URL: http://ion.ru